CLINICAL TRIAL: NCT04155788
Title: Food Exposure Therapy in Individuals With or Without Eating Disorders
Brief Title: Conquering Feared Foods Study
Acronym: CFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Cheri Levinson, Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 17.1288
Record Dates: First submitted 2019-09-16; First posted 2019-11-07 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Eating Disorder Symptom; Fear
Keywords: eating disorder; food exposure; feared food
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food Exposure (Experimental)
  Interventions: Behavioral: Food Exposure

INTERVENTIONS:
Behavioral: Food Exposure — Participants will complete a meal exposure using one of their feared foods.

SUMMARY:
The purpose of this study is to use ecological momentary assessment (EMA) data and physiological data to asses a client's eating disorder symptoms and behaviors before and after a meal with a feared food. The investigators are conducting a pilot clinical measurement study. Participants will be screened for eating disorder symptoms via a structured clinical interview. Participants with or without eating disorders will also complete self-reported measures of eating disorder symptoms and anxiety. Participants with eating disorders will complete assessments on their phone and will wear a sensor band to assess heart rate and galvanic skin response.

DETAILED DESCRIPTION:
Exposure therapy has been used in the treatment of Anorexia Nervosa (AN), as seen in mirror exposure to address body image and anxiety, as well as food exposure to address avoidant eating behavior. In food exposure therapy, individuals are exposed to feared foods in a clinical and/or non-clinical setting. Food exposure therapy has been effective in alleviating some anxiety in individuals with eating disorder behaviors and symptoms. However, the investigators do not yet know what characteristics predict response in food exposure therapy. The purpose of this study is to use EMA data and physiological data to asses a client's eating disorder symptoms and behaviors before and after a meal with a feared food.

Lastly, the study would like to utilize individuals who do not meet criteria for an eating disorder (ED) and will act as controls in this study to address the research question: is there a difference between individuals with EDs and without EDs as they complete the entirety of the study, specifically in regards to physiological data? These controls will not complete the EMA data aspect of the study.

The investigators are conducting a pilot clinical measurement study. Participants will be screened for eating disorder symptoms via a structured clinical interview or determined to not have eating disorder symptoms and will act as controls in the study. Both groups will also complete self-reported measures of eating disorder symptoms and anxiety. Participants will also complete assessments on their phone and will wear a sensor band to assess heart rate and galvanic skin response. However, control participants will not complete assessments on their phone. Both groups will wear the health-sensor band to assess heart rate and galvanic skin response.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 13-65, must meet criteria for a current diagnosis of anorexia nervosa or bulimia nervosa.
* Must be local to the Louisville area or able to travel to the study location for the two lab sessions.
* For participants to be in the control group, participants must be between the ages of 13-65.
* Must be local to the Louisville area or able to travel to the study location for the two lab sessions

Exclusion Criteria:

* Participants who are younger than 13 or older than 65 at the time of enrollment.
* Participants who are not local or can not travel to the Louisville area for the two therapy sessions.
* We will also exclude anyone who is actively suicidal (e.g., has a suicide plan), psychotic, or manic.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Self Reported Anxiety | through study completion, an average of four weeks
  Changes in Subjective Units of Distress Scale (SUDS) Ratings. The SUDS measures subjective units of distress on a scale from 0-100 where 0 indicates no anxiety and 100 indicates the most anxiety one has ever felt or could imagine feeling.
Physiological Data | through study completion, an average of four weeks
  Changes in heart rate
Participants' self-reported Safety Behaviors | through study completion, an average of four weeks
  Changes in behaviors done to alleviate anxiety as reported via open-ended questions about mealtimes. Prior to the study, participants are provided a brief training to understand common safety behaviors in eating disorders. Then, throughout the food exposure, they are periodically asked to identify any safety behaviors they are currently engaging in.

SECONDARY OUTCOMES:
Eating Disorder Symptoms & Behaviors | through study completion, an average of four weeks
  Changes in eating disordered symptoms and behaviors will be measured using a meal measure which identifies strategies used to avoid feelings of anxiety during meals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson HB, Wetterneck CT, Cahill SP, Steinglass JE, Franklin ME, Leonard RC, Weltzin TE, Riemann BC. Treatment of obsessive-compulsive disorder complicated by comorbid eating disorders. Cogn Behav Ther. 2013;42(1):64-76. doi: 10.1080/16506073.2012.751124. Epub 2013 Jan 15. PMID 23316878
- See also: Laboratory Website Description of Study — http://www.louisvilleeatlab.com/conquering-fear-foods-study.html